CLINICAL TRIAL: NCT02067793
Title: Phase 2, Randomized, Double-Blind, Multiple-Dose Level, Placebo Controlled, Single Intravenous Dose, Parallel Efficacy and Safety Study of NRX-1074 in Subjects With Major Depressive Disorder
Brief Title: Study of Intravenous NRX-1074 in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRX1074-C-201
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-02

CONDITIONS: Major Depressive Disorder
Keywords: NRX-1074; NMDA Receptor Modulator; Major Depressive Disorder; Glycine site modulator
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- NRX-1074 1 mg (Experimental): NRX-1074 1 mg, intravenous
  Interventions: Drug: NRX-1074 1 mg
- NRX-1074 5 mg (Experimental): NRX-1074 5 mg, intravenous
  Interventions: Drug: NRX-1074 5 mg
- NRX-1074 10 mg (Experimental): NRX-1074 10 mg, intravenous
  Interventions: Drug: NRX-1074 10 mg

INTERVENTIONS:
Drug: NRX-1074 1 mg — Single intravenous administration of 1 mg into arm on Day 0
  Other Names: NRX-1074 IV single dose
  Arms: NRX-1074 1 mg
Drug: Placebo — Single intravenous injection into the arm on Day 0
  Other Names: NRX-1074 IV single dose
  Arms: Placebo
Drug: NRX-1074 5 mg — Single intravenous injection of 5 mg into the arm on Day 0
  Other Names: NRX-1074 IV single dose
  Arms: NRX-1074 5 mg
Drug: NRX-1074 10 mg — Single intravenous injection of 10 mg into the arm on Day 0
  Other Names: NRX-1074 IV single dose
  Arms: NRX-1074 10 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of NRX-1074 following a single intravenous dose in subjects with major depressive disorder.

DETAILED DESCRIPTION:
NRX-1074 is a N-methyl-D-aspartate (NMDA) receptor functional partial agonist with efficacy in animal models of affective disorders including major depressive disorder. The purpose of this study is to evaluate efficacy and safety of NRX-1074 at dose levels that are predicted by comparison of human and animal pharmacokinetics to be efficacious.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* Aged 18 to 65 years
* Meets Diagnostic and Statistical Manual, Fourth Edition, Text Revision (DSM-IV-TR) criteria for major depressive disorder (MDD)
* Current episode has lasted ≥ 8 weeks before Screening
* HDRS-17 score ≥ 21 before beginning the washout of all current antidepressant agents and/or adjuvant agents
* HDRS-17 score ≥ 21 at Baseline (after 14 days of washout of current antidepressant agents)
* Female subjects of childbearing potential with a negative serum pregnancy test prior to entry into the study and who are practicing an adequate method of birth control (eg oral or parenteral contraceptives, intrauterine device, barrier, abstinence) and who do not plan to become pregnant during the course of the study. Female subjects may be included without a negative serum pregnancy test if they are surgically sterile or at least 2 years post-menopausal
* Male subjects and their female sexual partner should use an acceptable method of birth control during the study
* Clinical laboratory values < 2 times the upper limit of normal (ULN) or deemed not clinically significant per the investigator and Naurex medical monitor
* Ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments
* Based on both the investigator and Naurex medical monitor's clinical judgment, subjects with eating disorders, obsessive compulsive disorder (OCD), panic disorder, post-traumatic stress disorder (PTSD), and generalized anxiety disorders secondary to major depressive episodes are permitted

Exclusion Criteria:

* Axis I diagnosis of delirium, dementia, dysthymia, amnestic or other cognitive disorder, schizophrenia or other psychotic disorder, bipolar I or II disorder, eating disorder (anorexia or bulimia nervosa), obsessive-compulsive disorder, panic disorder, agoraphobia, social phobia, attention-deficit hyperactivity disorder (ADHD), or PTSD
* A clinically significant current Axis II diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal, or histrionic personality disorder
* Experiencing hallucinations, delusions, or any psychotic symptomatology in the current episode; lifetime history of psychosis
* Huntington's, Parkinson's, Alzheimer's, Multiple Sclerosis, or a history of seizures or strokes
* Currently hospitalized or residing in an in-patient facility during the study participation
* Substance abuse within the last 12 months, including greater than or equal to 5 units of alcohol per day where 1 unit = 1/2 pint of beer, 1 glass of wine, or 1 oz. of spirits consumed most weeks or in the opinion of the investigator
* Allergy or intolerance to current antidepressant or other current medications
* Participation in any clinical trial of an investigational product or device within 30 days of enrollment in this trial
* Positive screen for drugs of abuse: cocaine, marijuana, PCP, ketamine, opioid or other agent that in the opinion of the investigator is being abused
* Have received electroconvulsive therapy, transcranial magnetic stimulation (TMS), or vagal nerve stimulation (VNS) for the current depressive episode
* Post current (past 6 months) suicide risk based on administration of the C-SSRS and the investigator's clinical judgment
* Human immunodeficiency virus (HIV) infection (based on the HIV-1 & HIV-2 antibody screen) or other ongoing infectious disease
* Females or female partners of male subjects who are currently pregnant or planning to become pregnant during the course of the study. Women who are breastfeeding
* Currently taking prescription (psychiatric treatments, antidepressant treatments) or over-the-counter medications including herbal therapies to treat their MDD or conditions secondary to their period following study drug dosing. Dextromethorphan or tramadol since these are serotonin uptake inhibitors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the mean change from baseline in Hamilton Depression Rating Scale 17 (HDRS-17) score for each NRX-1074 dose group versus the placebo group's mean change | Day 1, Day 3, Day 7, Day 14
  Change in Hamilton Depression Rating Scale HDRS-17

SECONDARY OUTCOMES:
Change in Brief Psychiatric Rating Scale positive symptoms (BPRS+) scale | Day 1
Change in Clinician Administered Dissociative States Scale (CADSS) | Day 1
Change in Columbia-Suicide Severity Rating Scale (C-SSRS) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Naurex, Inc, an affiliate of Allergan plc
Locations (12):
- United States (12):
  - Pacific Research Partners, Oakland, California
  - Psychiatric Medicine Associates, Skokie, Illinois
  - University of Kansas School of Medicine Clinical Trial Unit, Wichita, Kansas
  - Boston Clinical Trials, Inc., Roslindale, Massachusetts
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - Mount Sinai School of Medicine, Elmsford, New York
  - New York State Psychiatric Institute, New York, New York
  - Lindner Center of HOPE, Mason, Ohio
  - Research Strategies Memphis, Memphis, Tennessee
  - Research Across America, Dallas, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Psychiatric Alliance of the Blue Ridge, Charlottesville, Virginia